CLINICAL TRIAL: NCT00800527
Title: Phase 4 Study of Efficacy of Gabapentin in the Treatment of Chest Pain and Paresthesia in Patients With Sternotomy
Brief Title: Efficacy of Gabapentin in the Treatment of Chest Pain and Paresthesia in Patients With Sternotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Usak State Hospital (Other)
Responsible Party: Ismail BIYIK, Investigator
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4ISM4350015-009/295
Record Dates: First submitted 2008-11-28; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Chest Pain; Paresthesia
Keywords: sternotomy; pain; paresthesia; Poststernotomy chest pain; Poststernotomy chest paresthesia
MeSH Terms: conditions — Chest Pain; Paresthesia; Pain | interventions — Gabapentin; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Gabapentin
  Interventions: Drug: Gabapentin
- 2 (Active Comparator): Diclofenac
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 800 mg one a day up to 30 day
  Other Names: Group-1: Gabapentin Arm
  Arms: 1
Drug: Diclofenac — Diclofenac 75 mg one a day up to 30 day
  Other Names: Group-2: Diclofenac arm
  Arms: 2

SUMMARY:
In this study, the investigators aim to demonstrate the efficacy of gabapentin compared with diclofenac in the treatment of chronic non-ischemic chest pain and paresthesia of the patients with sternotomy and to elucidate the similarities of PCPP to neuropathic pain syndromes.

DETAILED DESCRIPTION:
Because the primary objective of this study is to evaluate the effect of different drugs on chest pain and paresthesia, we choose the prospective, randomized, open label, blinded end point design for this study. According to this design, both patients and physicians making first assessment are aware of the treatment but the investigators making second and third assessment are blinded to treatment. Therefore, two separate cardiovascular surgeons wil select and randomize the patients and a cardiologist blinded to treatment assignments will evaluate the patients at second interview at thirty day and 3 months later. The study was approved by the Local Ethics Committee and informed consent was obtained from each patient. The study was conducted in Usak State Hospital with collaboration the Department of Cardiology of Ataturk Education and Training Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Poststernotomy chest pain and/or paresthesia

Exclusion Criteria:

* Osteoporosis, renal function impairment (creatinine value >1.5 mg / dl.)
* Hepatic dysfunction, peptic ulcer, chest pain with ischemic origin, pediatric cases
* Over production of scar tissue, thoracic surgery other than sternotomy -
* Redo-bypass surgery, infection, sternal dehiscence,valve surgery together with bypass

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Reduction of pain or paresthesia severity | one month

SECONDARY OUTCOMES:
duration of relief of pain or paresthesia | three month

CONTACTS AND LOCATIONS:
Overall Officials: Ismail BIYIK, MD, Principal Investigator — Investigator
Locations (1):
- Usak State Hospital, Uşak, Turkey (Türkiye)